CLINICAL TRIAL: NCT04150198
Title: MECHANISMS OF NEURONAL RESILIENCE IN ALZHEIMER'S DISEASE AND ITS FOCAL VARIANTS: A PET/MR STUDY
Acronym: PET-AL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: France Alzheimer (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: C19-40
Record Dates: First submitted 2019-10-22; First posted 2019-11-04 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease, Early Onset; Posterior Cortical Atrophy
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Nombre de participants 45 sujets répartis dans 3 groupes:
  1. Groupe MA-J (Maladie d'Alzheimer précoce)= 15 patients avec un diagnostic de MA-J
  2. Groupe ACP (Atrophie Corticale Posterieure)= 15 patients avec un diagnostic d'ACP
  3. Groupe sujets contrôles= 15 sujets contrôles
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with Alzheimer (<65 years) (AD-Y) (Experimental): 15 patients with a diagnostic of MA-J
  Interventions: Device: TEP/IRM
- Patients with posterior Cortical Atrophy (PCA) (Experimental): 15 patients with a diagnostic of PCA
  Interventions: Device: TEP/IRM
- Control (Active Comparator): 15 controls
  Interventions: Device: TEP/IRM

INTERVENTIONS:
Device: TEP/IRM — All participants will have a PET / MRI examination including: i) a 30-minute PET scan, 80 minutes after intravenous injection of 240 MBq of 18F-AV1451 ± 10% ii) a ZTE sequence (for attenuation correction of PET images), a 3D T1 anatomical sequence, a diffusion MRI, a functional MRI at rest (total duration: 45 minutes). These acquisitions will be made during the same exam session on a hybrid PET / MRI camera allowing simultaneous acquisitions. This visit lasts about 3 hours.

SUMMARY:
Patients with Alzheimer's disease and with early onset of symptoms (<65 years) (AD-Y) have a multi-domain cognitive deficit, whereas memory disorders (typical of the elderly patient's AD) are less often in the foreground. In addition, some MA-J have an atypical phenotype indicating focal brain damage, although they have the same pathological lesions: amyloid deposits and tau protein deposition (DNF). This is the case of posterior cortical atrophy (PCA) characterized by complex visual disturbances and atrophy affecting the more posterior regions of the brain. Based on the clinical profile of PCA patients, a more refined anatomo-clinical classification was proposed, distinguishing a rather "ventral" form and a rather "dorsal" form. The recent arrival of tau-specific PET tracers now makes it possible to evaluate in vivo fibrillary neurodegeneration (FND), which is well correlated with the severity of cognitive disorders. Advances in MRI have shown that each neurodegenerative syndrome targets a large-scale neural network, which in turn shows a vulnerability for a specific biological disease. In the case of AD, the reason for such a difference in cognitive and anatomical impairment between patients with diffuse involvement and others with more focal involvement is not known. One possible explanation is the existence, in focal forms, of neuronal mechanisms that oppose vulnerability. These mechanisms may correspond to the so-called "resilience" phenomenon, defined as resistance to a neuropathological process by the ability to optimize cognitive performance via the efficient recruitment of neural networks. The mechanisms underlying resilience in neurodegeneration are unknown. Their identification is very important for the management and treatment of AD.

DETAILED DESCRIPTION:
Working hypotheses We hypothesize that "focal" patients (PCA) versus "diffuse" patients (AD-Y) have (i) less severe white matter involvement; (ii) effective reorganization of the functional brain networks; iii) pathologically, a different topography and lesion load.

This project has no redundancy with the work already done in our team and in other teams at the international level.

Expected benefits This study will highlight the neural mechanisms underlying resiliency in a group of AD patients who, although having the same disease, present with a very different clinical and cognitive profile. Demonstration of these specific mechanisms of resilience in the diseased brain is essential to better understand the pathophysiological processes of AD. We consider that the pharmacological approach and the functional reeducation to this disease depend essentially on a better knowledge of both the topographic distribution of the underlying histopathology (in particular, the tau protein), and the response capacity from the brain to these lesions (state of connection of networks, functional reorganization). In addition, when treatments for AD are available, a precise definition of phenotypic variants will be essential for the selection of patients for these therapies and for therapeutic follow-up. In the longer term, resilient neural circuits could be modulated and strengthened through transcranial stimulation. Indeed, promising results have been obtained showing that these techniques can improve the performance of altered cognitive functions in patients with dementia.

ELIGIBILITY:
Inclusion Criteria:

1. For all subjects:

   * Affiliation to a social security insurance or beneficiary
   * Informed consent form signed by the participant or his / her legal representative
   * Participants aged 40 to 80 years.
2. Selection of AD-Y group

   - In vivo proof of Alzheimer's pathology:
   * Determination of specific proteins on the cerebrospinal fluid (CSF, a routine care procedure). The values considered pathological (AD) are Aβ1-42 peptide <500 (μg / ml), and / or tau protein> 450 and phosphorylated tau protein> 60, IATI index <1, tau / Aβ protein ratios > 1.23 as well as phosphorylated tau protein / Aβ1-42> 0.211.
   * And / or a positive PET-amyloid imaging test.
   * Early-onset episodic memory deficit (<65 years), progressive onset with evidence of hippocampal amnesic syndrome at neuropsychological assessment.

   In memory tests, the amnesic hippocampal syndrome is defined by: a deficit of the free recall despite a reinforced encoding, an effectiveness of the indexing or an impairment of the recognition capabilities, the presence of intrusions. The presence during the tests of false memories spontaneous (intrusions) or provoked (false recognitions) is also very contributive to the definition of amnesic syndrome of the hippocampal type.
3. PCA group selection

   Patients with a clinical and cognitive profile suggestive of PCA, characterized by:
   * an in vivo proof of the Alzheimer pathology (see selection of the AD-Y group)
   * a specific impairment of neuro-visual abilities, in the absence of major disorders of episodic memory (hippocampal) and executive functions.

   Two possible variants:
   * occipito-temporal variant: visuo-perceptive deficit in the foreground, early onset and progressive worsening; lack of visual identification of objects, symbols, words or faces;
   * biparietal variant: visuospatial deficit in the foreground, early settlement and progressive worsening; Gerstmann syndrome; Balint syndrome; gestural apraxia; visual-spatial neglect.
4. Selection of the control subjects group

   * Normal neurological and neuropsychological examinations.
   * Control subjects will be matched in age to patients.

Non-inclusion Criteria:

1. General non-inclusion criteria:

   * Medical history of torsade de pointe or risk of torsade de pointes
   * Patient treated with drugs known to lengthen QT (see www.crediblemeds.org)
   * Contraindication to radiopharmaceutical injection:

   For precautions of safety of use of the radiopharmaceutical, a blood sample allowing to check the renal and hepatic functions will be realized before imagery. The delay between the sampling and the neuroimaging visit is left to the investigator's discretion based on the patient's biological results. In particular, the glomerular filtration rate will be calculated from the results obtained.

   In the event of renal insufficiency (GFR 30mL / min / 1.73m2), hepatic insufficiency or any other biological anomaly of grade 3 or higher detected during these analyzes, the participant will not be able to carry out PET imaging. In this case, the results of the analyzes will be sent to the doctor indicated by the participant. This evaluation, which involves a determination of serum creatinine, is part of the standard routine biological assessment performed in the context of cognitive disorders

   Inability to provide informed consent by participant or legal representative:
   * Patient deprived of liberty by decision of justice or not benefiting from social cover.
   * Person in the process of participating in another therapeutic research or in a period of exclusion from another research.
   * Participants with a contraindication to MRI: pacemaker or cardiac defibrillator, implanted equipment activated by an electrical, magnetic or mechanical system, haemostatic clips of intracerebral aneurysms or carotid arteries , carriers of orthopedic implants.
   * Contraindication to radiopharmaceutical injection: known hypersensitivity to the active substance or to any of the excipients, renal impairment (GFR 30mL / min / 1.73m2), hepatic insufficiency or any other biological abnormality of grade 3 or higher
   * Person suffering from claustrophobia.
   * Pregnancy (for women of childbearing age, a urine pregnancy test will be performed on the day of the inclusion visit and the PET-MRI examination).
   * Any symptoms or biological values suggestive of a systemic disorder (renal, hepatic, cardiovascular, pulmonary) or any other medical conditions that could interfere with the interpretation of test results or compromise the health of patients.
   * Person subject to a legal safeguard.
2. Specific non-inclusion criteria for AD-Y and PCA patients:

   * Sudden appearance of cognitive deficits.
   * Gait disturbances, convulsions, major behavior modification.
   * Focal alterations to neurological examination, extrapyramidal signs, hallucinations, fluctuations. cognitive.
   * Psychiatric, cerebrovascular, metabolic, inflammatory pathology.
3. Specific non-inclusion criteria for control subjects:

   * Pathological neurological examination
   * History of neurological disease (in particular ischemic stroke or neurodegenerative disease) or psychiatric illness (particularly severe depression, psychosis, or bipolar illness still requiring drug treatment at the time of inclusion)
   * Physical affection that is serious or can interfere with cognitive functions.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
highlight of the "resilient" neural networks | up to 3 months
  For this, we will study:
  1) The topographic distribution regions of tau lesions, thanks to PET brain imaging using the 18F-AV-1451 as a ligand.
quantify the impairment (ie brain vulnerability) in AD-Y and in PCA | up to 3 months
  For this, we will study:
  2) The correlation between the distribution of these tau lesions and: the cortical volume, the indices of integrity of the white matter bundles, the functional neural networks, as well as the reorganization of the "hubs" of these networks, thanks to the structural MRI, diffusion (MRI) and functional at rest (fMRI) imaging.2)

SECONDARY OUTCOMES:
correlation between the concentration of tau-tauphosphorylated protein in cerebrospinal fluid (CSF) with the lesion load measured in PET | up to 3 months
  this comparison is a key element of characterization of this new ligand compared to widely validated CSF biomarkers
predictive model of functional alterations based on the structural alterations of the gray matter and the white matter. | up to 3 months
  To establish this correlation the evaluation criterion is represented by the measurement of cortical thickness, the indices of integrity of the beams of the white substance (fractional anisotropy, average, radial and perpendicular diffusivities), as well as the integration values of the functional networks and the distribution of "hubs"

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Service Hospitalier Frédéric Joliot SHFJ, Orsay
  - Service de Médecine Nucléaire - Hopital La Pitié Salpetriere, Paris

IPD SHARING:
Plan to Share IPD: Undecided